CLINICAL TRIAL: NCT03959800
Title: Genetic and Molecular Basis of Pediatric Liver Cancer
Brief Title: Molecular Basis of Pediatric Liver Cancer
Status: Recruiting | Type: Observational
Sponsor: University of Pittsburgh (Other)
Responsible Party: Principal Investigator, Rakesh Sindhi, Professor of Surgery, University of Pittsburgh
Other Study IDs: STUDY20050018
Record Dates: First submitted 2019-05-15; First posted 2019-05-22 (Actual); Last update posted 2025-09-12 (Actual); Status verified 2025-09

CONDITIONS: Childhood Liver Cancer; Liver Malignant Tumors; Embryonal Sarcoma of Liver (Disorder); Hepatoblastoma; Hepatocellular Carcinoma; Rhabdoid Tumor of Liver
Keywords: Hepatoblastoma; Hepatocellular Carcinoma; Pediatric Liver Cancer
MeSH Terms: conditions — Carcinoma, Hepatocellular; Hepatoblastoma

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Biospecimen Retention: Samples With DNA — Samples with DNA: blood, saliva or liver tissue.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The purpose of this retrospective and prospective project is to understand the molecular and genetic basis of liver cancer of childhood. Understanding the molecular and genetic bases of liver cancers can offer a better classification based on tumor biology, mechanisms and predisposition.

DETAILED DESCRIPTION:
Pediatric liver cancers are rare, affecting at times no more than 1 in one million population. Understanding the molecular basis of these cancers is important in order to develop more accurate diagnoses and more effective treatments. Current classifications of these cancers are based on how these cancers look on diagnostic studies such as radiologic imaging or under the microscope. Such a classification system does not explain why a particular cancer has a different outcome from what is considered "usual" for that particular cancer. Nor does such a classification system explain why two different classes of cancers behave the same way. Understanding the genetic bases of liver cancers can offer a better classification based on tumor biology, mechanisms and predisposition.

To achieve these goals, large numbers of such cancer patients or affected tissue must be collected. This is not possible in any single institution, or any single country. The current project will collect biological samples such as residual tumor tissue, saliva, or blood from affected patients and their biological parents and families, along with clinical information about the cancer. These biological samples will be used to study the genes and how these genes work in tumor tissue and in non-tumor tissue. The results of this study will permit childhood liver cancers to be categorized on the basis of common defects in genes and their function.

ELIGIBILITY:
Inclusion Criteria:

* Prior or current treatment for a childhood liver tumor, malignant or benign, at age <21 years.
* Biological parents and siblings of eligible children.

Exclusion Criteria:

* No prior or current treatment for a childhood liver tumor.
* Non-biological parents, legal guardians, or non-biological siblings of eligible children.

Ages: 0 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Living or deceased individuals who were diagnosed with a liver tumor, malignant or benign, during childhood (age <21 years) and their biological parents and siblings.
Sampling Method: Non-Probability Sample
Enrollment: 1600 (Estimated)
Dates: Start 2015-06-22 (Actual); Primary Completion 2028-06-30 (Estimated); Study Completion 2029-06-30 (Estimated)

PRIMARY OUTCOMES:
Gene sequencing | Recurrence free survival at 2 years
  DNA sequence variants
Gene expression analysis | Recurrence free survival at 2 years
  Differentially expressed genes
Status of genome-wide chromatin accessibility | Duration of active chemotherapy to two years after surgical treatment
  chromatin accessibility
Epigenetic change | Duration of active chemotherapy to two years after surgical treatment
  Differential methylation
Tumor infiltrating cells which express immune checkpoints | Duration of active chemotherapy to two years after surgical treatment
  differentially enriched immune cells

SECONDARY OUTCOMES:
Response to chemotherapy | Duration of active chemotherapy to two years after surgical treatment
  Survival
Response to chemotherapy | Duration of active chemotherapy to two years after surgical treatment
  Relapse

CONTACTS AND LOCATIONS:
Locations (1):
- UPMC Children's Hospital of Pittsburgh, Pittsburgh, Pennsylvania, United States